CLINICAL TRIAL: NCT03300596
Title: Suicidal Adults With Alcohol or Drug Use Problems: A New Hospital-based Treatment
Brief Title: Brief New Treatment for Suicide Attempts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kenneth Conner, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSRB00069554
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Suicide, Attempted; Drug Use; Alcohol; Use, Problem
MeSH Terms: conditions — Suicide, Attempted; Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- brief intervention to prevent suicide attempt (Experimental): Individuals presenting to hospital following a suicide attempt who are age 18-plus and screen positive for alcohol or drug use problem
  Interventions: Behavioral: Brief intervention to prevent suicide attempt
- standard of care (Other): Individuals presenting to hospital following a suicide attempt who are age 18-plus and screen positive for alcohol or drug use problem
  Interventions: Behavioral: Enhanced treatment as usual

INTERVENTIONS:
Behavioral: Brief intervention to prevent suicide attempt — A patient-centered, 3-session intervention that calls for videotaping the narrative story of a patient's suicide attempt, in his/her own words (session 1); reviewing segments of the tape to arrive at a shared understanding of the attempt and the sequence of events that led to it (session 2); and using this information, along with a homework task completed by the patient in-between sessions, in order to develop a collaborative, comprehensive written safety plan that addresses the patient's unique vulnerabilities (session 3).
  Other Names: Modification of the Attempted Suicide Short Intervention Program (ASSIP)
  Arms: brief intervention to prevent suicide attempt
Behavioral: Enhanced treatment as usual — Safety procedures' control intervention. For these procedures we will share summary results of the research assessments regarding suicidal thoughts, suicidal behaviors, alcohol and drug use and related problems, and depressive symptoms with appropriate hospital clinical staff. We will also arrange to send this information, with participants' permission, to their ongoing therapist or treatment program and, if none exists, to the therapist or program to which they are being referred. In this regard, the research assessment protocol serves a dual function of helping with additional monitoring of high-risk patients in addition to providing data for the study.
  Arms: standard of care

SUMMARY:
Individuals with alcohol or drug use problems who are hospitalized for suicide attempt are at high risk for reattempt. This treatment development study adapts a promising outpatient intervention to prevent suicide reattempt in order to administer it during hospitalization to individuals with alcohol and drug use problems, and to test the adapted intervention in a pilot randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* suicide attempt within one week of hospitalization with acknowledgment of some intent to die using a standard item
* problematic alcohol or drug use as determined by score >8 on Alcohol Use Disorders Identification Test, AUDIT or >3 on the 10-item version of the Drug Abuse Screening Test, DAST-10
* admission to hospital
* residence within 40 miles of Strong Memorial Hospital

Exclusion Criteria:

* under age 18
* treated in ED, CPEP, or observation unit only
* unable to communicate with the researcher in English
* unable to comprehend the nature of the study
* participation untenable from a medical (e.g., intubated), psychiatric (e.g., florid psychosis), or behavioral (e.g., refusing to speak with staff) standpoint
* short hospital length of stay, ruling out administering three sessions of the therapy prior to discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
suicide reattempt | 6 months
  number who reattempt suicide

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Conner KR, Kearns JC, Denneson LM. Qualitative analysis of hospital patient narratives of warning signs on the day of their suicide attempt. Gen Hosp Psychiatry. 2022 Nov-Dec;79:146-151. doi: 10.1016/j.genhosppsych.2022.11.001. Epub 2022 Nov 9. PMID 36375343
- [Derived] Conner KR, Kearns JC, Esposito EC, Pizzarello E, Wiegand TJ, Britton PC, Michel K, Gysin-Maillart AC, Goldston DB. Pilot RCT of the Attempted Suicide Short Intervention Program (ASSIP) adapted for rapid delivery during hospitalization to adult suicide attempt patients with substance use problems. Gen Hosp Psychiatry. 2021 Sep-Oct;72:66-72. doi: 10.1016/j.genhosppsych.2021.07.002. Epub 2021 Jul 19. PMID 34304029
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617